CLINICAL TRIAL: NCT03275285
Title: Randomized, Open Label, Multicenter Study Assessing The Clinical Benefit Of Isatuximab Combined With Carfilzomib (Kyprolis®) And Dexamethasone Versus Carfilzomib With Dexamethasone In Patients With Relapse And/Or Refractory Multiple Myeloma Previously Treated With 1 to 3 Prior Lines
Brief Title: Multinational Clinical Study Comparing Isatuximab, Carfilzomib And Dexamethasone To Carfilzomib And Dexamethasone In Relapse And/Or Refractory Multiple Myeloma Patients
Acronym: IKEMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EFC15246; U1111-1195-5957 (Registry Identifier: ICTRP); 2017-001940-37 (EudraCT Number)
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Results first posted 2023-02-13 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Plasma Cell Myeloma
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; carfilzomib; Dexamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Isatuximab + Carfilzomib + Dexamethasone (IKd) (Experimental): Isatuximab (intravenous) on day 1, 8, 15 and 22 of 1st cycle, then on day 1 and 15 of subsequent cycles in combination with carfilzomib (intravenous) on day 1, 2, 8, 9, 15 and 16 + dexamethasone (intravenous or by mouth [po]) on day 1, 2, 8, 9, 15, 16, 22 and 23 of a 28 day cycle.
  Interventions: Drug: isatuximab SAR650984; Drug: carfilzomib; Drug: dexamethasone
- Carfilzomib + Dexamethasone (Kd) (Active Comparator): Carfilzomib (intravenous) on day 1, 2, 8, 9, 15, 16 + dexamethasone (intravenous or po) on day 1, 2, 8, 9, 15, 16, 22 and 23 of a 28 day cycle.
  Interventions: Drug: carfilzomib; Drug: dexamethasone

INTERVENTIONS:
Drug: isatuximab SAR650984 — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Other Names: Sarclisa
  Arms: Isatuximab + Carfilzomib + Dexamethasone (IKd)
Drug: carfilzomib — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Other Names: Kyprolis
Drug: dexamethasone — Pharmaceutical form: tablets or solution for infusion
  Route of administration: oral or intravenous

SUMMARY:
The purpose of this study it to compare the efficacity of isatuximab when combined to carfilzomib and dexamethasone versus carfilzomib and dexamethasone in patients with multiple myeloma already treated with 1 to 3 prior lines of therapy.

DETAILED DESCRIPTION:
The duration of the study for a patient will include a period for screening of up to 3 weeks. Patients will be treated until disease progression, unacceptable AE, or patient decision to stop the study treatment. After study treatment discontinuation, patients will have follow-up visits until the analysis of overall survival.

ELIGIBILITY:
Inclusion criteria:

* Participants with MM previously treated with prior 1 to 3 lines and with measurable serum M-protein (>= 0.5 gram/deciliter) and/or urine M-protein (>= 200 milligram/24 hours).

Exclusion criteria:

* Participants previously pretreated with carfilzomib, who never achieved at least one minor response during previous therapies and/or last previous therapy completed within 14 last days.
* Participants with serum free light chain (FLC) measurable disease only.
* Participants less than 18 years old, participants with Eastern Cooperative Oncology Group performance status more than 2.
* Participants with inadequate biological tests.
* Participants with myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association class III or IV congestive heart failure, superior or equal to grade 3 arrhythmias, stroke or transient ischemic attack within last 6 months, and/or left ventricular ejection fraction lower than 40%.
* Participants with previous cancer unless disease free for more than 5 years or in situ cancer curatively treated.
* Participants with known acquired immunodeficiency syndrome related illness or human immunodeficiency virus requiring antiretroviral treatment, or hepatitis A, B, or C active infection.
* Women of childbearing potential or male participant with women of childbearing potential who do not agree to use highly effective method of birth control.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2025-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (70):
- United States (2):
  - UCSF MS Center Site Number : 8400002, San Francisco, California
  - Spartanburg Medical Center Site Number : 8400003, Spartanburg, South Carolina
- Australia (7):
  - Investigational Site Number : 0360005, Blacktown, New South Wales
  - Investigational Site Number : 0360006, Tweed Heads, New South Wales
  - Investigational Site Number : 0360002, Wollongong, New South Wales
  - Investigational Site Number : 0360001, Fitzroy, Victoria
  - Investigational Site Number : 0360004, Heidelberg West, Victoria
  - Investigational Site Number : 0360007, Nedlands, Western Australia
  - Investigational Site Number : 0360008, West Perth, Western Australia
- Brazil (5):
  - Hospital Sao Rafael - Rede D'OR Sao Luiz Site Number : 0760005, Salvador, Estado de Bahia
  - Hospital Mae de Deus Site Number : 0760003, Porto Alegre, Rio Grande do Sul
  - Hospital de Amor - Hospital do Cancer de Barretos - Fundacao Pio XII Site Number : 0760001, Barretos, São Paulo
  - Hospital das Clinicas de Sao Paulo Site Number : 0760002, São Paulo, São Paulo
  - Instituto COI de Educacao e Pesquisa Site Number : 0760004, Rio de Janeiro
- Canada (3):
  - Investigational Site Number : 1240003, Surrey, British Columbia
  - Investigational Site Number : 1240001, Saint John, New Brunswick
  - Investigational Site Number : 1240002, Montreal, Quebec
- Czechia (4):
  - Investigational Site Number : 2030002, Brno
  - Investigational Site Number : 2030004, Olomouc
  - Investigational Site Number : 2030003, Ostrava - Poruba
  - Investigational Site Number : 2030001, Prague
- France (6):
  - Investigational Site Number : 2500003, Lille
  - Investigational Site Number : 2500001, Nantes
  - Investigational Site Number : 2500006, Paris
  - Investigational Site Number : 2500002, Pessac
  - Investigational Site Number : 2500005, Pierre-Bénite
  - Investigational Site Number : 2500004, Poitiers
- Greece (5):
  - Investigational Site Number : 3000002, Athens
  - Investigational Site Number : 3000005, Athens
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000004, Pátrai
  - Investigational Site Number : 3000003, Thessaloniki
- Hungary (4):
  - Investigational Site Number : 3480003, Budapest
  - Investigational Site Number : 3480001, Budapest
  - Investigational Site Number : 3480004, Budapest
  - Investigational Site Number : 3480005, Kaposvár
- Italy (4):
  - Investigational Site Number : 3800003, Bologna
  - Investigational Site Number : 3800001, Pisa
  - Investigational Site Number : 3800004, Reggio Emilia
  - Investigational Site Number : 3800002, Torino
- Japan (7):
  - Investigational Site Number : 3920005, Shiwa-gun, Iwate
  - Investigational Site Number : 3920007, Kumamoto, Kumamoto
  - Investigational Site Number : 3920001, Suwa-shi, Nagano
  - Investigational Site Number : 3920003, Sunto-gun, Shizuoka
  - Investigational Site Number : 3920004, Shibuya-ku, Tokyo
  - Investigational Site Number : 3920006, Shinjuku-ku, Tokyo
  - Investigational Site Number : 3920002, Yamagata
- New Zealand (2):
  - Investigational Site Number : 5540001, Auckland
  - Investigational Site Number : 5540002, Wellington
- Russia (3):
  - Investigational Site Number : 6430003, Kirov
  - Investigational Site Number : 6430004, Novosibirsk
  - Investigational Site Number : 6430002, Yekaterinburg
- South Korea (5):
  - Investigational Site Number : 4100006, Busan, Busan
  - Investigational Site Number : 4100002, Gangnam-gu, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100005, Seoul
- Spain (5):
  - Investigational Site Number : 7240001, Badalona, Catalunya [Cataluña]
  - Investigational Site Number : 7240005, Barcelona, Catalunya [Cataluña]
  - Investigational Site Number : 7240002, Valencia, Valenciana, Comunidad
  - Investigational Site Number : 7240003, Madrid
  - Investigational Site Number : 7240004, Seville
- Turkey (Türkiye) (5):
  - Investigational Site Number : 7920003, Adana
  - Investigational Site Number : 7920001, Ankara
  - Investigational Site Number : 7920005, Bursa
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920004, Samsun
- United Kingdom (3):
  - Investigational Site Number : 8260004, Plymouth, Devon
  - Investigational Site Number : 8260005, Leicester, Leicestershire
  - Investigational Site Number : 8260001, Bristol, Somerset

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Moreau P, Dimopoulos MA, Mikhael J, Yong K, Capra M, Facon T, Hajek R, Spicka I, Baker R, Kim K, Martinez G, Min CK, Pour L, Leleu X, Oriol A, Koh Y, Suzuki K, Risse ML, Asset G, Mace S, Martin T; IKEMA study group. Isatuximab, carfilzomib, and dexamethasone in relapsed multiple myeloma (IKEMA): a multicentre, open-label, randomised phase 3 trial. Lancet. 2021 Jun 19;397(10292):2361-2371. doi: 10.1016/S0140-6736(21)00592-4. Epub 2021 Jun 4. PMID 34097854
- [Result] Martin TG, Capra M, Mohty M, Suzuki K, Quach H, Cavo M, Moreau P, Dimopoulos M, Yong K, Tekle C, Foster MC, Barnes Y, Risse ML, Mikhael J. Isatuximab Plus Carfilzomib and Dexamethasone Versus Carfilzomib and Dexamethasone in Patients with Relapsed Multiple Myeloma: IKEMA Subgroup Analysis by Prior Transplantation. Transplant Cell Ther. 2023 Feb;29(2):134.e1-134.e7. doi: 10.1016/j.jtct.2022.11.005. Epub 2022 Nov 11. PMID 36372355
- [Result] Chami B, Okuda M, Moayeri M, Pirenne F, Hidaka Y, Nambiar A, Song Z, Bedel O, Zhang B, Hopke J, Deng G, Zhu C, Mace S, Chiron M, Adrian F, Fukao T, Basile FG, Martin T. Anti-CD38 monoclonal antibody interference with blood compatibility testing: Differentiating isatuximab and daratumumab via functional epitope mapping. Transfusion. 2022 Nov;62(11):2334-2348. doi: 10.1111/trf.17137. Epub 2022 Oct 14. PMID 36239134
- [Derived] Yong K, Martin T, Dimopoulos MA, Mikhael J, Capra M, Facon T, Hajek R, Spicka I, Baker R, Kim K, Martinez G, Min CK, Pour L, Leleu X, Oriol A, Koh Y, Suzuki K, Casca F, Mace S, Risse ML, Moreau P. Isatuximab plus carfilzomib-dexamethasone versus carfilzomib-dexamethasone in patients with relapsed multiple myeloma (IKEMA): overall survival analysis of a phase 3, randomised, controlled trial. Lancet Haematol. 2024 Oct;11(10):e741-e750. doi: 10.1016/S2352-3026(24)00148-0. Epub 2024 Jul 24. PMID 39067465
- [Derived] Thoren K, Menad S, Nouadje G, Mace S. Isatuximab-Specific Immunofixation Electrophoresis Assay to Remove Interference in Serum M-Protein Measurement in Patients with Multiple Myeloma. J Appl Lab Med. 2024 Jul 1;9(4):661-671. doi: 10.1093/jalm/jfae028. PMID 38573925
- [Derived] Facon T, Moreau P, Baker R, Min CK, Leleu X, Mohty M, Karlin L, Armstrong NM, Tekle C, Schwab S, Risse ML, Martin T. Isatuximab plus carfilzomib and dexamethasone in patients with early versus late relapsed multiple myeloma: IKEMA subgroup analysis. Haematologica. 2024 Feb 1;109(2):604-616. doi: 10.3324/haematol.2023.283073. PMID 37584290
- [Derived] Kawano Y, Kim K, Min CK, Koh Y, Ishizawa K, Kim SH, Ito S, Tanaka J, Uchiyama M, Ishida T, Kim JS, Moreau P, Martin T, Tada K, Risse ML, Suzuki K. Isatuximab Plus Carfilzomib and Dexamethasone in East Asian Patients With Relapsed Multiple Myeloma: Updated IKEMA Subgroup Analysis. Clin Lymphoma Myeloma Leuk. 2023 Oct;23(10):e360-e367. doi: 10.1016/j.clml.2023.06.011. Epub 2023 Jul 3. PMID 37479547
- [Derived] Martin T, Dimopoulos MA, Mikhael J, Yong K, Capra M, Facon T, Hajek R, Spicka I, Baker R, Kim K, Martinez G, Min CK, Pour L, Leleu X, Oriol A, Koh Y, Suzuki K, Casca F, Mace S, Risse ML, Moreau P. Isatuximab, carfilzomib, and dexamethasone in patients with relapsed multiple myeloma: updated results from IKEMA, a randomized Phase 3 study. Blood Cancer J. 2023 May 9;13(1):72. doi: 10.1038/s41408-023-00797-8. PMID 37156782
- [Derived] Beksac M, Spicka I, Hajek R, Bringhen S, Jelinek T, Martin T, Mikala G, Moreau P, Symeonidis A, Rawlings AM, van de Velde H, Richardson PG. Evaluation of isatuximab in patients with soft-tissue plasmacytomas: An analysis from ICARIA-MM and IKEMA. Leuk Res. 2022 Nov;122:106948. doi: 10.1016/j.leukres.2022.106948. Epub 2022 Sep 6. PMID 36108425
- [Derived] Moreau P, Dimopoulos MA, Yong K, Mikhael J, Risse ML, Asset G, Martin T. Isatuximab plus carfilzomib/dexamethasone versus carfilzomib/dexamethasone in patients with relapsed/refractory multiple myeloma: IKEMA Phase III study design. Future Oncol. 2020 Jan;16(2):4347-4358. doi: 10.2217/fon-2019-0431. Epub 2019 Dec 13. PMID 31833394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 69 active centers in 16 countries. A total of 341 participants were screened between 25 October 2017 and 21 March 2019, of which 39 participants were screen failure due to not meeting eligibility criteria. Randomization was stratified by number of prior lines (1 versus >1) & revised international staging system (R-ISS) I or II versus III versus not classified. Reason for not completed = Reason for definitive treatment discontinuation.
Pre-assignment Details: First result analysis (A) reported was for a data cut-off date of 7 Feb 2020 for efficacy outcomes, 14 Jan 2022 for CR, MRD and PFS2. PFS data was reported at both cut-off dates: 7 Feb 2020 & 14 Jan 2022. Primary A of PFS refers to planned interim A conducted at 103 events (death/PD) with cut-off date 7 Feb 2020 & Final A of PFS conducted at 159 events with cut-off date 14 Jan 2022. Data cut-off for overall survival and LPLV was 7 Feb 2023 and 3 Jan 2025, respectively.
Groups:
- Carfilzomib + Dexamethasone (Kd): Participants received carfilzomib 20 milligrams per meter square (mg/m^2), intravenous (IV) infusion on Days 1, and 2 in Cycle 1, and then escalated to 56 mg/m^2 on Days 8, 9, 15 and 16 of Cycle 1 and then on Days 1, 2, 8, 9, 15 and 16 of each subsequent 28-day treatment cycle along with dexamethasone 20 milligrams (mg), orally (PO) or IV on Days 1, 2, 8, 9, 15, 16, 22 and 23 of each 28-day treatment cycle until disease progression or unacceptable adverse event or participant's decision to discontinue the study treatment or any other reason, whichever comes first (maximum exposure: 349 weeks).
- Isatuximab + Carfilzomib + Dexamethasone (IKd): Participants received isatuximab 10 milligrams per kilogram (mg/kg), IV infusion on Days 1, 8, 15 and 22 in Cycle 1, and then on Days 1 and 15 of each 28-day treatment cycle plus carfilzomib 20 mg/m^2, IV on Days 1, and 2 in Cycle 1, and then escalated to 56 mg/m^2 on Days 8, 9, 15 and 16 of Cycle 1 and then on Days 1, 2, 8, 9, 15 and 16 of each subsequent 28-day treatment cycle and dexamethasone 20 mg, PO or IV on Day 1, 2, 8, 9, 15, 16, 22 and 23 of each 28-day treatment cycle until disease progression or unacceptable adverse event or participant's decision to discontinue the study treatment or any other reason, whichever comes first (maximum exposure: 356 weeks).
Period: Overall Study
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Started | 123 | 179
Treated | 122 | 177
Completed | 0 | 0
Not Completed | 123 | 179
Not completed — Adverse Event | 24 | 29
Not completed — Progressive disease | 68 | 86
Not completed — Withdrawal by Subject | 18 | 21
Not completed — Treatment extension study | 1 | 24
Not completed — Randomized and not treated | 1 | 2
Not completed — Study discontinuation | 1 | 5
Not completed — Others | 10 | 12

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population.
Groups:
- Carfilzomib + Dexamethasone (Kd): Participants received carfilzomib 20 mg/m^2, IV infusion on Days 1, and 2 in Cycle 1, and then escalated to 56 mg/m^2 on Days 8, 9, 15 and 16 of Cycle 1 and then on Days 1, 2, 8, 9, 15 and 16 of each subsequent 28-day treatment cycle along with dexamethasone 20 mg, PO or IV on Days 1, 2, 8, 9, 15, 16, 22 and 23 of each 28-day treatment cycle until disease progression or unacceptable adverse event or participant's decision to discontinue the study treatment or any other reason, whichever comes first (maximum exposure: 349 weeks).
- Isatuximab + Carfilzomib + Dexamethasone (IKd): Participants received isatuximab 10 mg/kg, IV infusion on Days 1, 8, 15 and 22 in Cycle 1, and then on Days 1 and 15 of each 28-day treatment cycle plus carfilzomib 20 mg/m^2, IV on Days 1, and 2 in Cycle 1, and then escalated to 56 mg/m^2 on Days 8, 9, 15 and 16 of Cycle 1 and then on Days 1, 2, 8, 9, 15 and 16 of each subsequent 28-day treatment cycle and dexamethasone 20 mg, PO or IV on Day 1, 2, 8, 9, 15, 16, 22 and 23 of each 28-day treatment cycle until disease progression or unacceptable adverse event or participant's decision to discontinue the study treatment or any other reason, whichever comes first (maximum exposure: 356 weeks).
- Total: Total of all reporting groups
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd) | Total
Number analyzed (Participants) | 123 | 179 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (10.0) | 63.3 (9.8) | 63.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 78 | 133
  Male | 68 | 101 | 169
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 24 | 26 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 83 | 131 | 214
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 12 | 14 | 26

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With Overall Response (OR) as Determined by Independent Response Committee: Primary Analysis
Description: OR: participants with sCR, CR, VGPR & partial response (PR) as best overall response assessed by IRC using IMWG response criteria (from start of treatment until disease progression, death, initiation of further anti-myeloma treatment/cutoff date, whichever occurs 1st). sCR: negative immunofixation on serum & urine, disappearance of soft tissue plasmacytoma, <5% plasma cells in bone marrow aspirate (BMA) + normal FLC ratio (0.26-1.65), absence of clonal cells in bone marrow biopsy. CR: negative immunofixation on serum & urine, disappearance of soft tissue plasmacytoma, <5% plasma cells in BMA. VGPR: serum & urine M-protein detectable by immunofixation, not on electrophoresis/,>=90% reduction in serum M-protein + urine M-protein level <100mg/24h/,>=90% decrease in SPD compared to baseline in soft tissue plasmacytoma. PR:>=50% reduction of serum M-protein & decrease in 24h urinary M-protein by >=90%/<200mg/24h, if present at baseline,>=50% decrease in SPD of soft tissue plasmacytoma.
Time Frame: From randomization until the primary analysis data cut-off date of 7 Feb 2020 (the median duration of follow-up was 20.73 months)
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Groups:
- Carfilzomib + Dexamethasone (Kd): Participants received carfilzomib 20 mg/m^2, IV infusion on Days 1, and 2 in Cycle 1, and then escalated to 56 mg/m^2 on Days 8, 9, 15 and 16 of Cycle 1 and then on Days 1, 2, 8, 9, 15 and 16 of each subsequent 28-day treatment cycle along with dexamethasone 20 mg, PO or IV on Days 1, 2, 8, 9, 15, 16, 22 and 23 of each 28-day treatment cycle until disease progression or unacceptable adverse event or participant's decision to discontinue the study treatment or any other reason, whichever comes first (maximum exposure: 114 weeks).
- Isatuximab + Carfilzomib + Dexamethasone (IKd): Participants received isatuximab 10 mg/kg, IV infusion on Days 1, 8, 15 and 22 in Cycle 1, and then on Days 1 and Day 15 of each 28-day treatment cycle plus carfilzomib 20 mg/m^2, IV on Days 1, and 2 in Cycle 1, and then escalated to 56 mg/m^2 on Days 8, 9, 15 and 16 of Cycle 1 and then on Days 1, 2, 8, 9, 15 and 16 of each subsequent 28-day treatment cycle and dexamethasone 20 mg, PO or IV on Day 1, 2, 8, 9, 15, 16, 22 and 23 of each 28-day treatment cycle until disease progression or unacceptable adverse event or participant's decision to discontinue the study treatment or any other reason, whichever comes first (maximum exposure: 111 weeks).
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
percentage of participants | 82.9 | 86.6
Statistical Analysis 1: Comparison: Carfilzomib + Dexamethasone (Kd) vs Isatuximab + Carfilzomib + Dexamethasone (IKd); Statistical analysis for comparison of Overall Response between the Kd and IKd arms based on primary analysis; Test type: Superiority — A closed test procedure was used to control the Type I error rate from the primary efficacy endpoints sequentially through the secondary efficacy endpoints. No further testing would be performed unless the significance level had been reached on PFS and testing on subsequent endpoints were continued only if the null hypothesis for the previously tested endpoint was rejected; p = 0.1930, Cochran-Mantel-Haenszel — One-sided p-value based on Stratified Cochran-Mantel-Haenszel test. Threshold for statistical significance level at 0.025; One sided p-value was stratified based on randomization factors according to IRT

2. Secondary Outcome: Percentage of Participants With Very Good Partial Response (VGPR) or Better as Determined by Independent Response Committee: Primary Analysis
Description: VGPR or better: defined as participants with sCR, CR and VGPR as the best overall response (defined as best response from start of treatment until disease progression, death, initiation of further anti-myeloma treatment or cut-off date whichever occurs first) as per IRC. As per IMWG response criteria: sCR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas, <5% plasma cells in BMAs plus normal FLC ratio (0.26-1.65), absence of clonal cells in bone marrow biopsy. CR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas, <5% plasma cells in BMAs. VGPR: serum and urine M-protein detectable by immunofixation, not on electrophoresis/,>=90% reduction in serum M-protein plus urine M-protein level <100mg/24h/,>=90% decrease in SPD compared to baseline in soft tissue plasmacytoma.
Time Frame: as for outcome 1
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
percentage of participants | 56.1 | 72.6

3. Secondary Outcome: Percentage of Participants With VGPR or Better With Minimal Residual Disease (MRD) Negativity: Primary Analysis
Description: Percentage of participants with sCR, CR and VGPR for whom MRD assessed by sequencing was negative at any time after first dose of study treatment. MRD was assessed centrally by next-generation sequencing in bone marrow aspiration samples from participants who achieve VGPR or better, to determine depth of response at molecular level. VGPR or better: percentage of participants with sCR, CR and VGPR. sCR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas, <5% plasma cells in BMAs plus normal FLC ratio (0.26-1.65), absence of clonal cells in bone marrow biopsy. CR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas, <5% plasma cells in BMAs. VGPR: serum and urine M-protein detectable by immunofixation, not on electrophoresis/,>=90% reduction in serum M-protein plus urine M-protein level <100mg/24h/,>=90% decrease in SPD compared to baseline in soft tissue plasmacytoma.
Time Frame: as for outcome 1
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
percentage of participants | 13.0 | 29.6

4. Secondary Outcome: Percentage of Participants With VGPR or Better With Minimal Residual Disease (MRD) Negativity: Final Analysis
Description: Percentage of participants with sCR, CR and VGPR for whom MRD assessed by sequencing was negative at any time after first dose of study treatment. MRD was assessed centrally by next-generation sequencing in BM aspiration samples from participants who achieve VGPR or better, to determine depth of response at molecular level. VGPR or better: percentage of participants with sCR, CR and VGPR. sCR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas, <5% plasma cells in bone marrow aspirates plus normal FLC ratio, absence of clonal cells in bone marrow biopsy. CR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas, <5% plasma cells in bone marrow aspirates. VGPR: serum and urine M-protein detectable by immunofixation, not on electrophoresis/,>=90% reduction in serum M-protein plus urine M-protein level <100mg/24h/,>=90% decrease in SPD compared to baseline in soft tissue plasmacytoma.
Time Frame: From randomization until the final analysis data cut-off date of 14 Jan 2022 (the median duration of follow-up was 43.96 months)
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Groups:
- Carfilzomib + Dexamethasone (Kd): Participants received carfilzomib 20 mg/m^2, IV infusion on Days 1, and 2 in Cycle 1, and then escalated to 56 mg/m^2 on Days 8, 9, 15 and 16 of Cycle 1 and then on Days 1, 2, 8, 9, 15 and 16 of each subsequent 28-day treatment cycle along with dexamethasone 20 mg, PO or IV on Days 1, 2, 8, 9, 15, 16, 22 and 23 of each 28-day treatment cycle until disease progression or unacceptable adverse event or participant's decision to discontinue the study treatment or any other reason, whichever comes first (maximum exposure: 208 weeks).
- Isatuximab + Carfilzomib + Dexamethasone (IKd): Participants received isatuximab 10 mg/kg, IV infusion on Days 1, 8, 15 and 22 in Cycle 1, and then on Days 1 and Day 15 of each 28-day treatment cycle plus carfilzomib 20 mg/m^2, IV on Days 1, and 2 in Cycle 1, and then escalated to 56 mg/m^2 on Days 8, 9, 15 and 16 of Cycle 1 and then on Days 1, 2, 8, 9, 15 and 16 of each subsequent 28-day treatment cycle and dexamethasone 20 mg, PO or IV on Day 1, 2, 8, 9, 15, 16, 22 and 23 of each 28-day treatment cycle until disease progression or unacceptable adverse event or participant's decision to discontinue the study treatment or any other reason, whichever comes first (maximum exposure: 215 weeks).
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
percentage of participants | 13.8 | 33.5

5. Secondary Outcome: Percentage of Participants With Complete Response (CR) as Per Independent Response Committee: Final Analysis
Description: Complete response was defined as the participants with sCR and CR. IMWG response criteria for sCR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas, <5% plasma cells in bone marrow aspirates plus normal free light chain (FLC) ratio (0.26-1.65), absence of clonal cells in bone marrow biopsy. CR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas, <5% plasma cells in bone marrow aspirates. Complete response at the time of the final analysis was assessed with hydrashift isatuximab immunofixation electrophoresis (IFE) assay, which separated immunoglobulin G (IgG) isatuximab from IgG M protein.
Time Frame: as for outcome 4
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
percentage of participants | 28.5 | 44.1

6. Secondary Outcome: Percentage of Participants With Complete Response With MRD Negativity: Final Analysis
Description: MRD negativity was defined as the percentage of participants for whom MRD was negative by next-generation sequencing at any timepoint after first dose of study treatment. Threshold for negativity is 10^-5. MRD status in a participant was negative if at least one result of the assessment was negative in the participant otherwise MRD was considered as positive (MRD status reported as positive, missing or unevaluable). CR: participants with sCR and CR. IMWG response criteria for sCR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas, <5% plasma cells in bone marrow aspirates plus normal FLC ratio (0.26-1.65), absence of clonal cells in bone marrow biopsy. CR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas, <5% plasma cells in bone marrow aspirates. Complete response at the time of the final analysis was assessed with Hydrashift isatuximab IFE assay, which separated IgG isatuximab from IgG M protein.
Time Frame: as for outcome 4
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
percentage of participants | 12.2 | 26.3

7. Secondary Outcome: Overall Survival (OS)
Description: Overall survival, defined as the time from the date of randomization to death from any cause. The data reported is based on cut-off date of 7 Feb 2023.
Time Frame: From randomization until the final analysis data cut-off date of 7 Feb 2023 (the median duration of follow-up was 56.61 months)
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Carfilzomib + Dexamethasone (Kd): Participants received carfilzomib 20 mg/m^2, IV infusion on Days 1, and 2 in Cycle 1, and then escalated to 56 mg/m^2 on Days 8, 9, 15 and 16 of Cycle 1 and then on Days 1, 2, 8, 9, 15 and 16 of each subsequent 28-day treatment cycle along with dexamethasone 20 mg, PO or IV on Days 1, 2, 8, 9, 15, 16, 22 and 23 of each 28-day treatment cycle until disease progression or unacceptable adverse event or participant's decision to discontinue the study treatment or any other reason, whichever comes first (maximum exposure: 265 weeks).
- Isatuximab + Carfilzomib + Dexamethasone (IKd): Participants received isatuximab 10 mg/kg, IV infusion on Days 1, 8, 15 and 22 in Cycle 1, and then on Days 1 and Day 15 of each 28-day treatment cycle plus carfilzomib 20 mg/m^2, IV on Days 1, and 2 in Cycle 1, and then escalated to 56 mg/m^2 on Days 8, 9, 15 and 16 of Cycle 1 and then on Days 1, 2, 8, 9, 15 and 16 of each subsequent 28-day treatment cycle and dexamethasone 20 mg, PO or IV on Day 1, 2, 8, 9, 15, 16, 22 and 23 of each 28-day treatment cycle until disease progression or unacceptable adverse event or participant's decision to discontinue the study treatment or any other reason, whichever comes first (maximum exposure: 268 weeks).
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
months | 50.60 [38.932 to NA] — Upper limit of the confidence interval could not be reached due to less number of participants with the events. | NA [52.172 to NA] — Median value and the upper and lower limit of the confidence interval could not be calculated because of less than 50% of the participants had OS events.

8. Secondary Outcome: Duration of Response (DOR): Primary Analysis
Description: DOR: time (in months) from date of 1st IRC determined response for participants achieving PR/better to date of 1st documented PD determined by IRC/death, whichever happens 1st. If disease progression/death before analysis cut-off date was not observed, DOR was censored at date of last valid disease assessment performed prior to initiation of further anti-myeloma treatment/data cut-off date, whichever was 1st. PD (IMWG criteria): inc of >=25% from lowest confirmed value in any 1 of following criteria: serum M-protein (absolute inc must be >=0.5 g/dL), serum M-protein inc >=1g/dL if lowest M component was >=5g/dL; urine M-component (absolute inc must be >=200mg/24 hour),appearance of new lesion(s), >=50% inc from nadir in SPD of >1 lesion, or >=50% inc in the longest diameter of previous lesion >1 cm in short axis. PR: >=50% reduction of serum M-protein & reduction in 24h urinary M-protein by >=90%/<200mg/24 h. Estimated by Kaplan Meier method.
Time Frame: as for outcome 1
Population: Analysis was performed on the subset of participants with PR or better (defined as responders) in ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 102 | 155
months | NA [14.752 to NA] — Median and upper limit of confidence interval could not be calculated because of less than 50% of the participants reaching PR or better with PFS events (PFS events includes progression and death without progression). | NA [NA to NA] — Median and the upper and lower limit of confidence interval could not be calculated because of less than 50% of the participants reaching PR or better with PFS events (PFS events includes progression and death without progression).
Statistical Analysis 1: Comparison: Carfilzomib + Dexamethasone (Kd) vs Isatuximab + Carfilzomib + Dexamethasone (IKd); Test type: Superiority; Stratified Hazard Ratio = 0.425, 95% CI 2-sided [0.269 to 0.672] — Stratification was done on the number of prior lines of therapy (1 vs. >1) and R-ISS stage (I or II vs. III vs. not classified) according to IRT

9. Secondary Outcome: Time to Progression (TTP): Primary Analysis
Description: TTP was defined as time in months from randomization to the date of first documentation of PD (as determined by the IRC). If progression was not observed before the analysis cut-off date or the date of initiation of further anti-myeloma treatment, TTP was censored at the date of the last valid disease assessment not showing disease progression performed prior to initiation of a further anti-myeloma treatment (if any) or the analysis cut-off date, whichever comes first. As per IMWG criteria, PD was defined for participants with inc of >= 25% from lowest confirmed value in any one of the following criteria: serum M-protein (the absolute inc must be >= 0.5 g/dL), serum M-protein inc >=1 g/dL if the lowest M component was >=5 g/dL; urine M-component (the absolute inc must be >=200 mg/24hour), appearance of new lesion(s), >=50% inc from nadir in SPD of >1 lesion, or >=50% inc in the longest diameter of a previous lesion >1 centimeter in short axis.
Time Frame: as for outcome 1
Population: Analysis was performed on ITT population. Analysis was performed by Kaplan-Meier method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
months | 20.27 [16.986 to NA] — Upper limit of the confidence interval could not be reached due to less number of participants with the progression event. | NA [NA to NA] — Median and the upper and lower limit of confidence interval could not be calculated because of less than 50% of the participants with the progression event.
Statistical Analysis 1: Comparison: Carfilzomib + Dexamethasone (Kd) vs Isatuximab + Carfilzomib + Dexamethasone (IKd); Test type: Superiority; Stratified Hazard Ratio = 0.495, 95% CI 2-sided [0.324 to 0.757] — [estimate comment as in outcome 8, analysis 1]

10. Secondary Outcome: Time to First Response: Primary Analysis
Description: Time to first response was defined as the time (in months) from randomization to the date of first IRC determined response (PR or better) that is subsequently confirmed. In the absence of response, participants were censored at the earliest of the date of the last valid disease assessment before disease progression or death, the date of the last valid disease assessment before initiation of a further anti-myeloma treatment (if any) or the analysis cut-off date, whichever comes first. PR per IMWG criteria was defined as >=50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >=90% or to <200 mg/24 h. In addition to the above listed criteria, if present at baseline, a >=50% reduction in the size (SPD) of soft tissue plasmacytomas was also required.
Time Frame: as for outcome 1
Population: Analysis was performed on ITT population. Analysis was performed by Kaplan-Meier method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
months | 1.12 [1.051 to 1.183] | 1.08 [1.051 to 1.117]
Statistical Analysis 1: Comparison: Carfilzomib + Dexamethasone (Kd) vs Isatuximab + Carfilzomib + Dexamethasone (IKd); Test type: Superiority; Stratified Hazard Ratio = 1.143, 95% CI 2-sided [0.888 to 1.471]; Stratification was done on the number of prior lines of therapy (1 vs. >1) and R-ISS stage (I or II vs. III vs. not classified) according to IRT

11. Secondary Outcome: Time to Best Response: Primary Analysis
Description: Time to best response was defined as time (in months) from randomization to the date of first occurrence of IRC determined as best overall response (PR or better) that is subsequently confirmed. In absence of response, participants were censored at earliest date of last valid disease assessment before disease progression/death, date of last valid disease assessment before initiation of further anti-myeloma treatment (if any)/ analysis cut-off date, whichever was 1st. PR (IMWG criteria) was defined as >=50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >=90% or to <200 mg/24 h. In addition to above listed criteria, if present at baseline, a >=50% reduction in the size (SPD) of soft tissue plasmacytomas was also required. Best Overall Response was defined as the best response, using the IRC's assessment of response, from start of treatment until disease progression, death, initiation of further anti-myeloma treatment or cut-off date, whichever occurs 1st.
Time Frame: as for outcome 1
Population: Analysis was performed on ITT population. Analysis was performed by Kaplan-Meier method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
months | 3.78 [2.858 to 4.172] | 4.60 [3.811 to 5.257]
Statistical Analysis 1: Comparison: Carfilzomib + Dexamethasone (Kd) vs Isatuximab + Carfilzomib + Dexamethasone (IKd); Test type: Superiority; Stratified Hazard Ratio = 0.955, 95% CI 2-sided [0.740 to 1.233] — [estimate comment as in outcome 8, analysis 1]

12. Secondary Outcome: Second Progression Free Survival (PFS2): Final Analysis - Data Cut-off Date of 14 Jan 2022
Description: PFS2 defined as time (in months) from date of randomization to date of 1st documentation of PD (as assessed by investigator) after initiation of further anti-myeloma treatment /death from any cause, whichever comes 1st. Participants alive without progression after initiation of further anti-myeloma treatment before analysis cut-off date, PFS2 censored at date of last follow-up visit not showing disease progression after initiation of further anti-myeloma treatment /analysis cut-off date, whichever comes 1st. As per IMWG criteria, PD: defined for participants with increase of >= 25% from lowest confirmed value in any 1 of following criteria: serum M-protein (absolute increase must be >= 0.5 g/dL), serum M-protein increase >=1 g/dL if lowest M component was >=5 g/dL; urine M-component (absolute increase must be >=200 mg/24hour), appearance of new lesion(s), >=50% increase from nadir in SPD of >1 lesion, or >=50% increase in longest diameter of previous lesion >1 centimeter short axis.
Time Frame: as for outcome 4
Population: Analysis was performed on ITT population. Analysis was performed by Kaplan-Meier method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
months | 35.58 [24.049 to 40.509] | 47.18 [38.111 to NA] — Upper limit of confidence interval could not be calculated because not enough participants with PFS2 events.
Statistical Analysis 1: Comparison: Carfilzomib + Dexamethasone (Kd) vs Isatuximab + Carfilzomib + Dexamethasone (IKd); [Not specified]; Test type: Superiority — [Not specified]; [Stratified Hazard Ratio] = 0.683, 95% CI 2-sided [0.496 to 0.941] — [estimate comment as in outcome 8, analysis 1]

13. Secondary Outcome: Second Progression Free Survival (PFS2): Overal Survival Analysis - Data Cut-off Date of 07 Feb 2023
Description: as for outcome 12
Time Frame: From randomization until the overal survival analysis data cut-off date of 07 Feb 2023 (the median duration of follow-up was 56.61 months)
Population: Analysis was performed on ITT population. Analysis was performed by Kaplan-Meier method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
months | 32.36 [23.129 to 40.016] | 47.18 [38.965 to 57.922]
Statistical Analysis 1: Comparison: Carfilzomib + Dexamethasone (Kd) vs Isatuximab + Carfilzomib + Dexamethasone (IKd); [Not specified]; Test type: Superiority — [Not specified]; Stratified Hazard Ratio = 0.663, 95% CI 2-sided [0.491 to 0.895] — [estimate comment as in outcome 8, analysis 1]

14. Secondary Outcome: Number of Participants With Renal Response (RR): Primary Analysis
Description: RR comprises of complete RR (CR renal), partial RR (PR renal) & minor RR (MR renal). CR renal was defined as an improvement in estimated glomerular filtration rate (eGFR) from <50 mL/min/1.73m^2 at Baseline to >=60 mL/min/1.73m^2 in at least 1 assessment during the treatment period (time from first dose of study treatment up to 30 days after last dose of study treatment); PR renal was defined as improvement in eGFR from <15 mL/min/1.73m^2 at baseline to at least 1 assessment in the range of 30 to 60 mL/min/1.73m^2 during the on-treatment-period and MR renal was defined as an improvement in eGFR from <15 mL/min/1.73m^2 at Baseline to at least 1 assessment in the range of 15 to 30 mL/min/1.73m^2 during the on-treatment-period or from 15 to 30 mL/min/1.73m^2 at Baseline to at least 1 assessment in the range of 30 to 60 mL/min/1.73m^2 during the on-treatment-period.
Time Frame: From the first dose of study treatment to 30 days following the last administration of study treatment (maximum duration: up to 114 weeks)
Population: Analysis was performed on ITT population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'Number analyzed' signifies participants with available data for each specified category. Here, "0" signifies that none of the participants were available for assessment at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 13 | 25
Participants
  CR Renal | 4 | 13
  PR Renal: number analyzed (Participants) | 0 | 0
  MR Renal: number analyzed (Participants) | 3 | 4
  MR Renal | 1 | 4

15. Secondary Outcome: Health Related Quality of Life (HRQL): Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Cancer Specific Questionnaire With 30 Items (EORTC QLQ-C30): Global Health Status Score at Specified Timepoints
Description: EORTC QLQ-C30 is a cancer-specific instrument that contains 30 items & provides multidimensional assessment of HRQL. EORTC QLQ-C30 includes global health status/quality of life (GHS/QOL), functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, nausea/vomiting), and 6 single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, financial difficulties). Most questions from QLQ-C30 are 4-point scale (1/Not at All to 4/Very Much), except Items 29-30, which comprise GHS scale & are 7-point scale (1/Very Poor to 7/Excellent). GHS total score is calculated as ([{Q29+Q30}/2]-1)/6*100. Answers are converted into grading scale, with values between 0 (worse outcome) to100 (best outcome). High score represents a favorable outcome with best quality of life for participant. Results reported for primary analysis with data cut-off date 7-Feb-2020.
Time Frame: Baseline, Day 1 of each cycle (Cycle 2 to Cycle 25), at the End of Treatment visit (any day up to 114 weeks)
Population: Analysis was performed on ITT population. Here, 'Number analyzed' signifies participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
score on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 99 | 151
  Cycle 2 Day 1 | 1.52 (21.11) | -1.60 (20.06)
  Cycle 3 Day 1: number analyzed (Participants) | 100 | 154
  Cycle 3 Day 1 | 4.17 (22.92) | 0.05 (20.29)
  Cycle 4 Day 1: number analyzed (Participants) | 100 | 150
  Cycle 4 Day 1 | 3.58 (21.20) | -1.89 (23.71)
  Cycle 5 Day 1: number analyzed (Participants) | 95 | 149
  Cycle 5 Day 1 | 3.60 (21.80) | -1.23 (23.12)
  Cycle 6 Day 1: number analyzed (Participants) | 88 | 145
  Cycle 6 Day 1 | 3.13 (20.50) | -1.44 (22.12)
  Cycle 7 Day 1: number analyzed (Participants) | 85 | 141
  Cycle 7 Day 1 | 4.22 (22.55) | -1.77 (22.38)
  Cycle 8 Day 1: number analyzed (Participants) | 83 | 134
  Cycle 8 Day 1 | 3.82 (21.71) | -1.06 (20.78)
  Cycle 9 Day 1: number analyzed (Participants) | 77 | 128
  Cycle 9 Day 1 | 6.60 (19.28) | -0.78 (22.17)
  Cycle 10 Day 1: number analyzed (Participants) | 73 | 124
  Cycle 10 Day 1 | 4.91 (21.55) | -1.21 (20.35)
  Cycle 11 Day 1: number analyzed (Participants) | 71 | 121
  Cycle 11 Day 1 | 4.34 (20.06) | -1.10 (20.18)
  Cycle 12 Day 1: number analyzed (Participants) | 64 | 119
  Cycle 12 Day 1 | 8.59 (22.37) | 0.84 (22.40)
  Cycle 13 Day 1: number analyzed (Participants) | 60 | 112
  Cycle 13 Day 1 | 7.08 (19.76) | -1.26 (20.63)
  Cycle 14 Day 1: number analyzed (Participants) | 59 | 111
  Cycle 14 Day 1 | 9.75 (21.62) | -0.98 (21.43)
  Cycle 15 Day 1: number analyzed (Participants) | 57 | 103
  Cycle 15 Day 1 | 5.26 (22.14) | 0.16 (20.51)
  Cycle 16 Day 1: number analyzed (Participants) | 50 | 101
  Cycle 16 Day 1 | 6.33 (20.73) | -1.07 (20.94)
  Cycle 17 Day 1: number analyzed (Participants) | 47 | 99
  Cycle 17 Day 1 | 7.27 (21.04) | 0.00 (22.18)
  Cycle 18 Day 1: number analyzed (Participants) | 45 | 92
  Cycle 18 Day 1 | 8.70 (23.16) | -0.36 (20.56)
  Cycle 19 Day 1: number analyzed (Participants) | 41 | 88
  Cycle 19 Day 1 | 12.40 (21.42) | -1.23 (20.12)
  Cycle 20 Day 1: number analyzed (Participants) | 34 | 87
  Cycle 20 Day 1 | 10.78 (20.97) | -1.05 (20.40)
  Cycle 21 Day 1: number analyzed (Participants) | 28 | 72
  Cycle 21 Day 1 | 12.50 (21.81) | -1.85 (21.54)
  Cycle 22 Day 1: number analyzed (Participants) | 19 | 53
  Cycle 22 Day 1 | 17.98 (22.27) | 0.31 (21.24)
  Cycle 23 Day 1: number analyzed (Participants) | 15 | 37
  Cycle 23 Day 1 | 15.56 (22.02) | 3.15 (20.73)
  Cycle 24 Day 1: number analyzed (Participants) | 9 | 22
  Cycle 24 Day 1 | 14.81 (26.28) | 0.38 (14.88)
  Cycle 25 Day 1: number analyzed (Participants) | 5 | 16
  Cycle 25 Day 1 | 15.00 (28.50) | 3.13 (17.18)
  End of Treatment: number analyzed (Participants) | 57 | 56
  End of Treatment | -6.14 (22.90) | -11.90 (25.86)

16. Secondary Outcome: HRQL: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Cancer Specific Questionnaire With 20 Items (EORTC QLQ-MY20): Disease Symptoms Domain Score at Specified Timepoints: Primary Analysis
Description: EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in participants with multiple myeloma. It is used in conjunction with the EORTC QLQ-C30 to assess symptoms and side effects due to treatment or the disease. Disease symptoms domain is one of the four domain scores. Disease symptoms domain consist of 6 questions and the score uses 4-point scale (1 'Not at All' to 4 'Very Much'). Disease Symptoms Domain Score is calculated as ([{Q31+Q32+Q33+Q34+Q35+Q36}/6]-1)/3*100. Scores are averaged, and transformed to 0-100 scale, where higher scores = more symptoms and lower HRQL.
Time Frame: Baseline, Day 1 of each cycle (Cycle 2 to Cycle 25), at the End of Treatment visit (any day up to 114 weeks)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
score on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 103 | 157
  Cycle 2 Day 1 | -5.34 (15.75) | -3.40 (19.58)
  Cycle 3 Day 1: number analyzed (Participants) | 102 | 158
  Cycle 3 Day 1 | -8.28 (15.33) | -7.42 (18.15)
  Cycle 4 Day 1: number analyzed (Participants) | 102 | 152
  Cycle 4 Day 1 | -5.45 (17.48) | -7.46 (17.99)
  Cycle 5 Day 1: number analyzed (Participants) | 97 | 150
  Cycle 5 Day 1 | -5.78 (17.01) | -6.37 (18.32)
  Cycle 6 Day 1: number analyzed (Participants) | 91 | 146
  Cycle 6 Day 1 | -6.11 (18.07) | -6.16 (19.88)
  Cycle 7 Day 1: number analyzed (Participants) | 87 | 143
  Cycle 7 Day 1 | -6.64 (17.44) | -4.78 (20.77)
  Cycle 8 Day 1: number analyzed (Participants) | 84 | 136
  Cycle 8 Day 1 | -6.94 (17.76) | -5.47 (19.96)
  Cycle 9 Day 1: number analyzed (Participants) | 79 | 131
  Cycle 9 Day 1 | -5.65 (18.00) | -5.51 (17.86)
  Cycle 10 Day 1: number analyzed (Participants) | 74 | 125
  Cycle 10 Day 1 | -5.56 (18.48) | -4.98 (17.24)
  Cycle 11 Day 1: number analyzed (Participants) | 72 | 122
  Cycle 11 Day 1 | -3.24 (17.78) | -7.10 (17.57)
  Cycle 12 Day 1: number analyzed (Participants) | 65 | 121
  Cycle 12 Day 1 | -5.30 (16.27) | -6.89 (17.58)
  Cycle 13 Day 1: number analyzed (Participants) | 60 | 114
  Cycle 13 Day 1 | -7.69 (17.06) | -5.95 (16.44)
  Cycle 14 Day 1: number analyzed (Participants) | 59 | 113
  Cycle 14 Day 1 | -8.66 (16.35) | -7.08 (17.98)
  Cycle 15 Day 1: number analyzed (Participants) | 57 | 105
  Cycle 15 Day 1 | -5.56 (17.69) | -5.19 (17.84)
  Cycle 16 Day 1: number analyzed (Participants) | 51 | 102
  Cycle 16 Day 1 | -8.06 (18.27) | -5.77 (18.66)
  Cycle 17 Day 1: number analyzed (Participants) | 47 | 101
  Cycle 17 Day 1 | -7.57 (19.01) | -4.29 (19.73)
  Cycle 18 Day 1: number analyzed (Participants) | 45 | 94
  Cycle 18 Day 1 | -7.16 (17.67) | -3.78 (17.93)
  Cycle 19 Day 1: number analyzed (Participants) | 41 | 90
  Cycle 19 Day 1 | -7.18 (19.57) | -3.64 (16.70)
  Cycle 20 Day 1: number analyzed (Participants) | 34 | 88
  Cycle 20 Day 1 | -11.93 (17.09) | -3.54 (21.63)
  Cycle 21 Day 1: number analyzed (Participants) | 28 | 73
  Cycle 21 Day 1 | -9.72 (16.74) | -3.81 (19.70)
  Cycle 22 Day 1: number analyzed (Participants) | 19 | 54
  Cycle 22 Day 1 | -9.94 (18.76) | -5.35 (22.48)
  Cycle 23 Day 1: number analyzed (Participants) | 15 | 37
  Cycle 23 Day 1 | -5.56 (25.11) | -6.01 (19.53)
  Cycle 24 Day 1: number analyzed (Participants) | 9 | 22
  Cycle 24 Day 1 | -6.17 (29.97) | -9.60 (18.16)
  Cycle 25 Day 1: number analyzed (Participants) | 5 | 16
  Cycle 25 Day 1 | -12.22 (28.97) | -14.58 (21.65)
  End of Treatment: number analyzed (Participants) | 59 | 57
  End of Treatment | 2.35 (23.10) | 1.75 (23.48)

17. Secondary Outcome: HRQL: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Cancer Specific Questionnaire With 20 Items (EORTC QLQ-MY20): Side Effects of Treatment at Specified Timepoints: Primary Analysis
Description: EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in participants with multiple myeloma. Side effects of treatment domain is one of the four domain scores. Side effects of treatment domain consists of 10 questions and the score uses a 4-point scale (1 'Not at All' to 4 'Very Much'). Side Effects of Treatment Score (MYSE) is calculated as ([{Q37+Q38+Q39+Q40+Q41+Q42+Q43+Q44+Q45+Q46}/10]-1)/3*100. Scores are averaged, and transformed to 0-100 scale, where higher scores = more side effects and lower HRQL and lower scores = less side effects and better HRQL.
Time Frame: Baseline, Day 1 of each cycle (Cycle 2 to Cycle 25), at the End of Treatment visit (any day up to 114 weeks)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
score on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 103 | 157
  Cycle 2 Day 1 | 1.23 (11.56) | 1.41 (11.71)
  Cycle 3 Day 1: number analyzed (Participants) | 102 | 158
  Cycle 3 Day 1 | 0.44 (10.11) | 0.84 (12.00)
  Cycle 4 Day 1: number analyzed (Participants) | 102 | 152
  Cycle 4 Day 1 | 0.83 (11.38) | 0.99 (11.89)
  Cycle 5 Day 1: number analyzed (Participants) | 97 | 150
  Cycle 5 Day 1 | 1.91 (11.36) | 2.36 (11.94)
  Cycle 6 Day 1: number analyzed (Participants) | 91 | 146
  Cycle 6 Day 1 | 2.08 (11.81) | 1.61 (12.32)
  Cycle 7 Day 1: number analyzed (Participants) | 87 | 143
  Cycle 7 Day 1 | 1.47 (12.14) | 2.14 (10.76)
  Cycle 8 Day 1: number analyzed (Participants) | 84 | 136
  Cycle 8 Day 1 | 1.53 (12.07) | 2.86 (12.77)
  Cycle 9 Day 1: number analyzed (Participants) | 79 | 131
  Cycle 9 Day 1 | 1.68 (11.57) | 1.49 (11.96)
  Cycle 10 Day 1: number analyzed (Participants) | 74 | 125
  Cycle 10 Day 1 | 2.07 (11.62) | 2.68 (12.51)
  Cycle 11 Day 1: number analyzed (Participants) | 72 | 122
  Cycle 11 Day 1 | 3.38 (12.00) | 2.03 (12.16)
  Cycle 12 Day 1: number analyzed (Participants) | 65 | 121
  Cycle 12 Day 1 | 1.20 (10.52) | 3.04 (12.72)
  Cycle 13 Day 1: number analyzed (Participants) | 60 | 114
  Cycle 13 Day 1 | 0.82 (10.22) | 2.12 (12.33)
  Cycle 14 Day 1: number analyzed (Participants) | 59 | 113
  Cycle 14 Day 1 | 1.08 (10.56) | 1.71 (12.58)
  Cycle 15 Day 1: number analyzed (Participants) | 57 | 105
  Cycle 15 Day 1 | 1.85 (11.45) | 1.87 (11.80)
  Cycle 16 Day 1: number analyzed (Participants) | 51 | 102
  Cycle 16 Day 1 | 0.99 (10.54) | 2.58 (11.88)
  Cycle 17 Day 1: number analyzed (Participants) | 47 | 101
  Cycle 17 Day 1 | 2.74 (10.03) | 4.10 (12.77)
  Cycle 18 Day 1: number analyzed (Participants) | 45 | 94
  Cycle 18 Day 1 | 2.37 (10.51) | 2.95 (13.38)
  Cycle 19 Day 1: number analyzed (Participants) | 41 | 90
  Cycle 19 Day 1 | 2.76 (11.41) | 2.16 (11.56)
  Cycle 20 Day 1: number analyzed (Participants) | 34 | 88
  Cycle 20 Day 1 | -0.17 (10.62) | 2.05 (13.03)
  Cycle 21 Day 1: number analyzed (Participants) | 28 | 73
  Cycle 21 Day 1 | 3.17 (10.61) | 2.74 (12.87)
  Cycle 22 Day 1: number analyzed (Participants) | 19 | 54
  Cycle 22 Day 1 | 3.55 (6.46) | 1.51 (12.51)
  Cycle 23 Day 1: number analyzed (Participants) | 15 | 37
  Cycle 23 Day 1 | 7.85 (9.93) | -1.39 (12.02)
  Cycle 24 Day 1: number analyzed (Participants) | 9 | 22
  Cycle 24 Day 1 | 12.35 (7.17) | -2.54 (11.33)
  Cycle 25 Day 1: number analyzed (Participants) | 5 | 16
  Cycle 25 Day 1 | 11.85 (4.06) | -3.50 (12.83)
  End of Treatment: number analyzed (Participants) | 59 | 57
  End of Treatment | 4.63 (13.01) | 5.56 (16.22)

18. Secondary Outcome: HRQL: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Cancer Specific Questionnaire With 20 Items (EORTC QLQ-MY20): Body Image Score at Specified Timepoints: Primary Analysis
Description: EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in participants with multiple myeloma. It is used in conjunction with the EORTC QLQ-C30 to assess symptoms and side effects due to treatment or the disease. It consists of one question and scores are based on the 4-point Likert scale ranging from "Not at all" to "Very much". Body image score is calculated as: (1 - [Q47-1]/3)*100. Scores are averaged, and transformed to scale ranging from 0 to 100. A higher score represents a better quality of life.
Time Frame: Baseline, Day 1 of each cycle (Cycle 2 to Cycle 25), at the End of Treatment visit (any day up to 114 weeks)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
score on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 103 | 157
  Cycle 2 Day 1 | -1.29 (23.76) | -1.27 (21.31)
  Cycle 3 Day 1: number analyzed (Participants) | 101 | 158
  Cycle 3 Day 1 | 1.98 (23.01) | 1.27 (26.84)
  Cycle 4 Day 1: number analyzed (Participants) | 101 | 152
  Cycle 4 Day 1 | -1.65 (25.55) | -1.10 (28.04)
  Cycle 5 Day 1: number analyzed (Participants) | 97 | 150
  Cycle 5 Day 1 | -0.69 (26.34) | -2.89 (27.29)
  Cycle 6 Day 1: number analyzed (Participants) | 91 | 146
  Cycle 6 Day 1 | -1.83 (24.02) | -1.60 (26.93)
  Cycle 7 Day 1: number analyzed (Participants) | 87 | 143
  Cycle 7 Day 1 | -0.77 (27.83) | -3.03 (24.36)
  Cycle 8 Day 1: number analyzed (Participants) | 84 | 136
  Cycle 8 Day 1 | -5.16 (25.08) | -0.25 (24.84)
  Cycle 9 Day 1: number analyzed (Participants) | 78 | 131
  Cycle 9 Day 1 | -2.14 (24.82) | -1.02 (25.80)
  Cycle 10 Day 1: number analyzed (Participants) | 74 | 125
  Cycle 10 Day 1 | -1.80 (25.22) | -1.33 (25.54)
  Cycle 11 Day 1: number analyzed (Participants) | 72 | 122
  Cycle 11 Day 1 | -1.85 (29.01) | -0.55 (23.47)
  Cycle 12 Day 1: number analyzed (Participants) | 65 | 121
  Cycle 12 Day 1 | -2.05 (25.60) | -0.55 (25.09)
  Cycle 13 Day 1: number analyzed (Participants) | 60 | 114
  Cycle 13 Day 1 | -3.89 (26.10) | -2.63 (21.79)
  Cycle 14 Day 1: number analyzed (Participants) | 59 | 113
  Cycle 14 Day 1 | -4.52 (26.59) | -3.24 (25.57)
  Cycle 15 Day 1: number analyzed (Participants) | 57 | 105
  Cycle 15 Day 1 | 0.00 (25.20) | -2.22 (24.58)
  Cycle 16 Day 1: number analyzed (Participants) | 51 | 102
  Cycle 16 Day 1 | -1.31 (27.46) | -2.94 (22.55)
  Cycle 17 Day 1: number analyzed (Participants) | 47 | 101
  Cycle 17 Day 1 | -1.42 (28.62) | -1.98 (26.17)
  Cycle 18 Day 1: number analyzed (Participants) | 45 | 94
  Cycle 18 Day 1 | 1.48 (30.11) | -1.77 (24.62)
  Cycle 19 Day 1: number analyzed (Participants) | 41 | 90
  Cycle 19 Day 1 | 0.00 (31.62) | -3.70 (26.18)
  Cycle 20 Day 1: number analyzed (Participants) | 34 | 88
  Cycle 20 Day 1 | 0.00 (27.22) | -0.76 (24.75)
  Cycle 21 Day 1: number analyzed (Participants) | 28 | 73
  Cycle 21 Day 1 | -4.76 (34.80) | -3.20 (26.74)
  Cycle 22 Day 1: number analyzed (Participants) | 19 | 54
  Cycle 22 Day 1 | -8.77 (36.59) | -1.85 (27.02)
  Cycle 23 Day 1: number analyzed (Participants) | 15 | 37
  Cycle 23 Day 1 | -13.33 (30.34) | -5.41 (24.23)
  Cycle 24 Day 1: number analyzed (Participants) | 9 | 22
  Cycle 24 Day 1 | -25.93 (36.43) | -3.03 (25.01)
  Cycle 25 Day 1: number analyzed (Participants) | 5 | 16
  Cycle 25 Day 1 | -53.33 (18.26) | -8.33 (25.82)
  End of Treatment: number analyzed (Participants) | 59 | 57
  End of Treatment | -5.65 (21.58) | -9.36 (27.28)

19. Secondary Outcome: HRQL: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Cancer Specific Questionnaire With 20 Items (EORTC QLQ-MY20): Future Perspective at Specified Timepoints: Primary Analysis
Description: EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in participants with multiple myeloma. It is used in conjunction with the EORTC QLQ-C30 to assess symptoms and side effects due to treatment or the disease. It consists of three questions and the scores are based on the 4-point Likert scale ranging from "Not at all" to "Very much". Future Perspective score is calculated as (1 - ([{Q48+Q49+Q50}/3] -1)/3)*100. Scores are averaged and transformed to scale ranging from 0 to 100. A higher score represents a better quality of life.
Time Frame: Baseline, Day 1 of each cycle (Cycle 2 to Cycle 25), at the End of Treatment visit (any day up to 114 weeks)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
score on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 103 | 157
  Cycle 2 Day 1 | 0.54 (19.33) | 7.57 (26.48)
  Cycle 3 Day 1: number analyzed (Participants) | 101 | 158
  Cycle 3 Day 1 | 4.84 (22.08) | 9.70 (24.76)
  Cycle 4 Day 1: number analyzed (Participants) | 101 | 152
  Cycle 4 Day 1 | 6.60 (20.44) | 8.55 (26.62)
  Cycle 5 Day 1: number analyzed (Participants) | 97 | 150
  Cycle 5 Day 1 | 7.67 (22.64) | 7.56 (26.98)
  Cycle 6 Day 1: number analyzed (Participants) | 91 | 146
  Cycle 6 Day 1 | 8.42 (21.81) | 9.97 (25.70)
  Cycle 7 Day 1: number analyzed (Participants) | 87 | 143
  Cycle 7 Day 1 | 8.17 (21.93) | 8.47 (24.74)
  Cycle 8 Day 1: number analyzed (Participants) | 84 | 136
  Cycle 8 Day 1 | 7.41 (22.51) | 10.54 (24.50)
  Cycle 9 Day 1: number analyzed (Participants) | 78 | 131
  Cycle 9 Day 1 | 7.26 (21.10) | 8.57 (28.26)
  Cycle 10 Day 1: number analyzed (Participants) | 74 | 125
  Cycle 10 Day 1 | 8.56 (22.79) | 11.56 (24.82)
  Cycle 11 Day 1: number analyzed (Participants) | 72 | 122
  Cycle 11 Day 1 | 8.02 (21.69) | 12.02 (24.23)
  Cycle 12 Day 1: number analyzed (Participants) | 65 | 121
  Cycle 12 Day 1 | 6.84 (24.51) | 11.48 (22.90)
  Cycle 13 Day 1: number analyzed (Participants) | 60 | 114
  Cycle 13 Day 1 | 11.11 (20.04) | 10.72 (23.18)
  Cycle 14 Day 1: number analyzed (Participants) | 59 | 113
  Cycle 14 Day 1 | 8.85 (22.86) | 11.31 (23.29)
  Cycle 15 Day 1: number analyzed (Participants) | 57 | 105
  Cycle 15 Day 1 | 9.55 (24.16) | 12.28 (22.27)
  Cycle 16 Day 1: number analyzed (Participants) | 51 | 102
  Cycle 16 Day 1 | 12.42 (24.51) | 11.76 (25.20)
  Cycle 17 Day 1: number analyzed (Participants) | 47 | 101
  Cycle 17 Day 1 | 12.29 (21.64) | 10.89 (25.29)
  Cycle 18 Day 1: number analyzed (Participants) | 45 | 94
  Cycle 18 Day 1 | 11.36 (22.41) | 7.33 (23.25)
  Cycle 19 Day 1: number analyzed (Participants) | 41 | 90
  Cycle 19 Day 1 | 9.21 (24.96) | 8.40 (25.50)
  Cycle 20 Day 1: number analyzed (Participants) | 34 | 88
  Cycle 20 Day 1 | 10.13 (24.67) | 9.60 (25.34)
  Cycle 21 Day 1: number analyzed (Participants) | 28 | 73
  Cycle 21 Day 1 | 10.32 (22.41) | 10.65 (26.15)
  Cycle 22 Day 1: number analyzed (Participants) | 19 | 54
  Cycle 22 Day 1 | 8.77 (25.28) | 12.14 (22.35)
  Cycle 23 Day 1: number analyzed (Participants) | 15 | 37
  Cycle 23 Day 1 | 9.63 (27.81) | 12.61 (20.48)
  Cycle 24 Day 1: number analyzed (Participants) | 9 | 22
  Cycle 24 Day 1 | 1.23 (24.50) | 16.16 (18.70)
  Cycle 25 Day 1: number analyzed (Participants) | 5 | 16
  Cycle 25 Day 1 | -4.44 (24.34) | 15.28 (16.67)
  End of Treatment: number analyzed (Participants) | 59 | 57
  End of Treatment | -3.95 (22.86) | -3.70 (31.45)

20. Secondary Outcome: HRQL: Change From Baseline in European Quality of Life Group Questionnaire With 5 Dimensions and 5 Levels Per Dimension (EQ-5D-5L): Health State Utility Index Value at Specified Timepoints: Primary Analysis
Description: The EQ-5D-5L is a standardized measure of health status that provides a general assessment of health utility and consist in 2 sections a descriptive system comprising 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and Visual Analog Scale (VAS). Each dimension has a 5-level response: no problems, slight problems, moderate problems, severe problems, and extreme problems. Response options are measured with a 5-point Likert scale. The 5D-5L systems are converted into a single index utility score between 0 to 1, where higher score indicates a better health state and lower score indicate worse health state.
Time Frame: Baseline, Day 1 of each cycle (Cycle 2 to Cycle 25), at the End of Treatment visit (any day up to 114 weeks)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
score on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 99 | 151
  Cycle 2 Day 1 | 0.05 (0.17) | 0.04 (0.19)
  Cycle 3 Day 1: number analyzed (Participants) | 98 | 150
  Cycle 3 Day 1 | 0.06 (0.21) | 0.05 (0.22)
  Cycle 4 Day 1: number analyzed (Participants) | 99 | 147
  Cycle 4 Day 1 | 0.02 (0.21) | 0.05 (0.21)
  Cycle 5 Day 1: number analyzed (Participants) | 95 | 144
  Cycle 5 Day 1 | 0.04 (0.20) | 0.04 (0.20)
  Cycle 6 Day 1: number analyzed (Participants) | 88 | 141
  Cycle 6 Day 1 | 0.03 (0.19) | 0.05 (0.23)
  Cycle 7 Day 1: number analyzed (Participants) | 85 | 139
  Cycle 7 Day 1 | 0.06 (0.19) | 0.04 (0.21)
  Cycle 8 Day 1: number analyzed (Participants) | 81 | 132
  Cycle 8 Day 1 | 0.06 (0.19) | 0.05 (0.22)
  Cycle 9 Day 1: number analyzed (Participants) | 77 | 124
  Cycle 9 Day 1 | 0.05 (0.20) | 0.04 (0.19)
  Cycle 10 Day 1: number analyzed (Participants) | 71 | 120
  Cycle 10 Day 1 | 0.06 (0.22) | 0.03 (0.22)
  Cycle 11 Day 1: number analyzed (Participants) | 69 | 118
  Cycle 11 Day 1 | 0.04 (0.23) | 0.05 (0.20)
  Cycle 12 Day 1: number analyzed (Participants) | 63 | 115
  Cycle 12 Day 1 | 0.03 (0.16) | 0.02 (0.20)
  Cycle 13 Day 1: number analyzed (Participants) | 59 | 109
  Cycle 13 Day 1 | 0.06 (0.16) | 0.03 (0.19)
  Cycle 14 Day 1: number analyzed (Participants) | 58 | 109
  Cycle 14 Day 1 | 0.06 (0.24) | 0.04 (0.19)
  Cycle 15 Day 1: number analyzed (Participants) | 57 | 101
  Cycle 15 Day 1 | 0.05 (0.18) | 0.05 (0.18)
  Cycle 16 Day 1: number analyzed (Participants) | 50 | 98
  Cycle 16 Day 1 | 0.06 (0.16) | 0.04 (0.19)
  Cycle 17 Day 1: number analyzed (Participants) | 46 | 97
  Cycle 17 Day 1 | 0.05 (0.15) | 0.03 (0.20)
  Cycle 18 Day 1: number analyzed (Participants) | 45 | 90
  Cycle 18 Day 1 | 0.02 (0.15) | 0.04 (0.17)
  Cycle 19 Day 1: number analyzed (Participants) | 41 | 86
  Cycle 19 Day 1 | 0.03 (0.20) | 0.03 (0.18)
  Cycle 20 Day 1: number analyzed (Participants) | 34 | 85
  Cycle 20 Day 1 | 0.06 (0.17) | 0.03 (0.23)
  Cycle 21 Day 1: number analyzed (Participants) | 28 | 70
  Cycle 21 Day 1 | 0.03 (0.15) | 0.02 (0.22)
  Cycle 22 Day 1: number analyzed (Participants) | 19 | 52
  Cycle 22 Day 1 | 0.05 (0.19) | 0.02 (0.22)
  Cycle 23 Day 1: number analyzed (Participants) | 15 | 36
  Cycle 23 Day 1 | 0.05 (0.18) | 0.00 (0.27)
  Cycle 24 Day 1: number analyzed (Participants) | 9 | 22
  Cycle 24 Day 1 | 0.04 (0.24) | 0.03 (0.20)
  Cycle 25 Day 1: number analyzed (Participants) | 5 | 16
  Cycle 25 Day 1 | 0.05 (0.38) | 0.04 (0.22)
  End of Treatment: number analyzed (Participants) | 57 | 56
  End of Treatment | -0.03 (0.25) | -0.08 (0.27)

21. Secondary Outcome: HRQL: Change From Baseline in European Quality of Life Working Group Health Status Measure 5 Dimensions, 5 Levels (EQ-5D-5L) Score: Visual Analogic Scale (VAS) at Specified Timepoints: Primary Analysis
Description: The EQ-5D-5L is a standardized measure of health status that provides a general assessment of health utility and consist of 2 sections; descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and a VAS. The VAS records the respondent's self-rated health on a 20 centimeter (cm) vertical VAS; the scale went from 0 (worst imaginable health state) to 100 (best imaginable health state). This information can be used as a quantitative measure of health as judged by the individual respondents.
Time Frame: Baseline, Day 1 of each cycle (Cycle 2 to Cycle 25), at the End of Treatment visit (any day up to 114 weeks)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
score on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 99 | 151
  Cycle 2 Day 1 | 2.42 (17.04) | 0.60 (15.23)
  Cycle 3 Day 1: number analyzed (Participants) | 98 | 150
  Cycle 3 Day 1 | 4.70 (16.13) | 3.47 (17.80)
  Cycle 4 Day 1: number analyzed (Participants) | 99 | 147
  Cycle 4 Day 1 | 6.03 (16.73) | 2.29 (18.69)
  Cycle 5 Day 1: number analyzed (Participants) | 94 | 144
  Cycle 5 Day 1 | 3.40 (16.89) | 2.35 (19.73)
  Cycle 6 Day 1: number analyzed (Participants) | 88 | 141
  Cycle 6 Day 1 | 2.80 (18.56) | 1.24 (19.11)
  Cycle 7 Day 1: number analyzed (Participants) | 84 | 139
  Cycle 7 Day 1 | 0.64 (21.69) | 2.24 (18.85)
  Cycle 8 Day 1: number analyzed (Participants) | 81 | 132
  Cycle 8 Day 1 | 1.48 (17.11) | 2.40 (18.87)
  Cycle 9 Day 1: number analyzed (Participants) | 77 | 124
  Cycle 9 Day 1 | -0.14 (17.46) | 2.93 (19.04)
  Cycle 10 Day 1: number analyzed (Participants) | 71 | 120
  Cycle 10 Day 1 | 2.76 (17.41) | 2.82 (18.35)
  Cycle 11 Day 1: number analyzed (Participants) | 69 | 118
  Cycle 11 Day 1 | 3.86 (20.07) | 3.77 (18.51)
  Cycle 12 Day 1: number analyzed (Participants) | 63 | 115
  Cycle 12 Day 1 | 5.29 (18.51) | 3.63 (19.34)
  Cycle 13 Day 1: number analyzed (Participants) | 59 | 109
  Cycle 13 Day 1 | 6.81 (19.57) | 4.94 (18.41)
  Cycle 14 Day 1: number analyzed (Participants) | 58 | 109
  Cycle 14 Day 1 | 7.95 (18.12) | 4.72 (17.67)
  Cycle 15 Day 1: number analyzed (Participants) | 57 | 101
  Cycle 15 Day 1 | 4.96 (18.92) | 3.23 (18.87)
  Cycle 16 Day 1: number analyzed (Participants) | 50 | 98
  Cycle 16 Day 1 | 3.94 (18.78) | 4.56 (18.88)
  Cycle 17 Day 1: number analyzed (Participants) | 46 | 97
  Cycle 17 Day 1 | 5.04 (17.93) | 4.97 (18.55)
  Cycle 18 Day 1: number analyzed (Participants) | 45 | 90
  Cycle 18 Day 1 | 3.71 (19.08) | 3.83 (18.46)
  Cycle 19 Day 1: number analyzed (Participants) | 41 | 86
  Cycle 19 Day 1 | 7.44 (18.73) | 3.69 (18.37)
  Cycle 20 Day 1: number analyzed (Participants) | 34 | 85
  Cycle 20 Day 1 | 6.18 (18.43) | 4.20 (17.20)
  Cycle 21 Day 1: number analyzed (Participants) | 28 | 70
  Cycle 21 Day 1 | 7.25 (23.46) | 3.26 (18.97)
  Cycle 22 Day 1: number analyzed (Participants) | 19 | 52
  Cycle 22 Day 1 | 5.58 (24.06) | 2.35 (18.62)
  Cycle 23 Day 1: number analyzed (Participants) | 15 | 36
  Cycle 23 Day 1 | 6.33 (18.73) | 6.44 (18.34)
  Cycle 24 Day 1: number analyzed (Participants) | 9 | 22
  Cycle 24 Day 1 | 5.11 (17.93) | 4.50 (18.31)
  Cycle 25 Day 1: number analyzed (Participants) | 5 | 16
  Cycle 25 Day 1 | 9.20 (21.48) | 5.00 (18.83)
  End of Treatment: number analyzed (Participants) | 57 | 56
  End of Treatment | -4.40 (18.66) | -7.80 (21.08)

22. Secondary Outcome: Pharmacokinetics: Plasma Concentration at End of Infusion (Ceoi) of Isatuximab: Primary Analysis
Description: Ceoi is the plasma concentration observed at the end of intravenous infusion.
Time Frame: End of infusion on Cycle 1 Day 1 and Cycle 1 Day 15; Cycle 2 Day 1
Population: Analysis was performed on pharmacokinetic (PK) population which included participants who received at least 1 dose of Isatuximab, with data for at least 1 PK parameter available. Data for this outcome measure (OM) was not planned to be collected and analyzed for Kd arm. Here, 'Number analyzed' signifies participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: microgram/milliliter (mcg/mL)
Arm/Group | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 172
microgram/milliliter (mcg/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 169
  Cycle 1 Day 1 | 274.01 (183.67)
  Cycle 1 Day 15: number analyzed (Participants) | 27
  Cycle 1 Day 15 | 380.28 (85.70)
  Cycle 2 Day 1: number analyzed (Participants) | 161
  Cycle 2 Day 1 | 522.74 (204.11)

23. Secondary Outcome: Pharmacokinetics: Plasma Concentration of Isatuximab at Ctrough: Primary Analysis
Description: Ctrough was the plasma concentration observed just before treatment administration during repeated dosing.
Time Frame: Pre-infusion on Cycle 1 Day 1, Day 8, Day 15 and Day 22, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, Cycle 7 Day 1, Cycle 8 Day 1, Cycle 9 Day 1 and Cycle 10 Day 1
Population: Analysis was performed on PK population. Data for this OM was not planned to be collected and analyzed for Kd arm. Here,'Number analyzed' signifies participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 172
mcg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 166
  Cycle 1 Day 1 | 3.66 (34.40)
  Cycle 1 Day 8: number analyzed (Participants) | 152
  Cycle 1 Day 8 | 82.14 (43.87)
  Cycle 1 Day 15: number analyzed (Participants) | 144
  Cycle 1 Day 15 | 180.02 (71.83)
  Cycle 1 Day 22: number analyzed (Participants) | 147
  Cycle 1 Day 22 | 252.63 (100.16)
  Cycle 2 Day 1: number analyzed (Participants) | 130
  Cycle 2 Day 1 | 324.28 (132.98)
  Cycle 3 Day 1: number analyzed (Participants) | 145
  Cycle 3 Day 1 | 295.78 (146.11)
  Cycle 4 Day 1: number analyzed (Participants) | 137
  Cycle 4 Day 1 | 342.48 (140.94)
  Cycle 5 Day 1: number analyzed (Participants) | 135
  Cycle 5 Day 1 | 389.25 (172.11)
  Cycle 6 Day 1: number analyzed (Participants) | 130
  Cycle 6 Day 1 | 427.16 (188.51)
  Cycle 7 Day 1: number analyzed (Participants) | 123
  Cycle 7 Day 1 | 433.22 (177.11)
  Cycle 8 Day 1: number analyzed (Participants) | 118
  Cycle 8 Day 1 | 490.51 (198.17)
  Cycle 9 Day 1: number analyzed (Participants) | 113
  Cycle 9 Day 1 | 486.07 (181.34)
  Cycle 10 Day 1: number analyzed (Participants) | 100
  Cycle 10 Day 1 | 490.08 (206.53)

24. Secondary Outcome: Pharmacokinetics: Maximum Observed Concentration (Cmax) of Carfilzomib: Primary Analysis
Description: Cmax was defined as the maximum concentration observed after the first infusion calculated using the non-compartmental analysis after the intravenous infusion of carfilzomib with isatuximab.
Time Frame: Cycle 1: pre-dose (0 hour), 30 minutes (min), 35 min, 45 min, 60 min, 1 hour 30 min, 2 hours 30 min and 4 hours 30 min post-dose on Day 15
Population: Analysis was performed on PK population. Data for this OM was not planned to be collected and analyzed for Kd arm. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 16
nanogram/milliliter (ng/mL) | 2090 (1360)

25. Secondary Outcome: Pharmacokinetics: Clast of Carfilzomib: Primary Analysis
Description: Clast was defined as the last concentration observed above the lower limit of quantification.
Time Frame: Cycle 1: pre-dose (0 hour), 30 min, 35 min, 45 min, 60 min, 1 hour 30 min, 2 hours 30 min and 4 hours 30 min post-dose on Day 15
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 16
ng/mL | 3.00 (5.11)

26. Secondary Outcome: Pharmacokinetics: Tmax of Carfilzomib: Primary Analysis
Description: Tmax was defined as the time to reach Cmax, calculated using the non-compartmental analysis after the intravenous infusion of carfilzomib with isatuximab.
Time Frame: as for outcome 25
Population: as for outcome 24
Measure: Median (Full Range); unit: hours
Arm/Group | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 16
hours | 0.54 [0.35 to 0.75]

27. Secondary Outcome: Pharmacokinetics: Tlast of Carfilzomib: Primary Analysis
Description: Tlast was defined as the time of last concentration observed above the lower limit of quantification, calculated using the non-compartmental analysis after the intravenous infusion of carfilzomib with isatuximab.
Time Frame: as for outcome 25
Population: as for outcome 24
Measure: Median (Full Range); unit: hours
Arm/Group | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 16
hours | 4.50 [2.52 to 4.75]

28. Secondary Outcome: Pharmacokinetics: Area Under the Plasma Concentration Time Curve (AUC) of Carfilzomib: Primary Analysis
Description: AUC was defined as area under the plasma concentration-time curve extrapolated to infinity according to the equation: AUC= AUClast + Clast/λz. AUC was calculated using the non-compartmental analysis after the intravenous infusion of carfilzomib with isatuximab.
Time Frame: as for outcome 25
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: nanograms*hour/milliliter(ng*h/mL)
Arm/Group | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 16
nanograms*hour/milliliter(ng*h/mL) | 784 (509)

29. Secondary Outcome: Pharmacokinetics: Area Under the Plasma Concentration Time Curve From Time 0 to Last Quantifiable Concentration (AUClast) of Carfilzomib: Primary Analysis
Description: AUClast was defined as area under the plasma concentration versus time curve calculated from time 0 to last quantifiable concentration. AUClast was calculated using the non-compartmental analysis after the intravenous infusion of carfilzomib with isatuximab.
Time Frame: as for outcome 25
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 16
ng*h/mL | 779 (505)

30. Secondary Outcome: Pharmacokinetics: Percentage of Extrapolation of AUC (AUCext) of Carfilzomib: Primary Analysis
Description: AUCext was defined as the percentage of the extrapolation of AUC, calculated using the non-compartmental analysis after the intravenous infusion of carfilzomib with isatuximab.
Time Frame: as for outcome 25
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC
Arm/Group | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 16
percentage of AUC | 0 (172)

31. Secondary Outcome: Pharmacokinetics: Terminal Half-life (t1/2z) of Carfilzomib: Primary Analysis
Description: T1/2 was defined as the time required for the concentration of the drug to reach half of its original value, calculated using the non-compartmental analysis after the intravenous infusion of carfilzomib with isatuximab.
Time Frame: as for outcome 25
Population: as for outcome 24
Measure: Median (Full Range); unit: hours
Arm/Group | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 16
hours | 0.860 [0.450 to 1.89]

32. Secondary Outcome: Pharmacokinetics: Clearance at Steady State (CLss) of Carfilzomib: Primary Analysis
Description: CLss was defined as a quantitative measure of the rate at which a drug substance is removed from the body at steady state, calculated using the non-compartmental analysis after the intravenous infusion of carfilzomib with isatuximab.
Time Frame: as for outcome 25
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Liters/hour (L/h)
Arm/Group | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 16
Liters/hour (L/h) | 466 (1190)

33. Secondary Outcome: Pharmacokinetics: Volume of Distribution at Steady State (Vss) of Carfilzomib: Primary Analysis
Description: Volume of Distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vss is the apparent volume of distribution at steady-state, calculated using the non-compartmental analysis after the intravenous infusion of carfilzomib with isatuximab.
Time Frame: as for outcome 25
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 16
Liters | 453 (1570)

34. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA): Primary Analysis
Description: ADA were categorized as: pre-existing, treatment induced, and treatment boosted response. Pre-existing ADA was defined as ADA that were present in samples drawn during the pretreatment period (i.e., before the first isatuximab administration). Treatment-induced ADA was defined as ADA that developed at any time during the ADA on-study observation period in participants without pre-existing ADA, including participants without pretreatment samples. Treatment boosted ADA was defined as pre-existing ADA with an increase in titer during the ADA on-study observation period.
Time Frame: From first dose of study treatment up to 30 days after last dose of study treatment (maximum duration: 111 weeks)
Population: Analysis was performed on ADA evaluable population which included participants who received at least one dose of study drug from the IKd arm with at least one ADA assessment during the ADA on-study observation period with a reportable result. Data for this outcome measure was not planned to be collected and analyzed for Kd arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 168
Participants
  Pre-existing ADA | 0
  Treatment induced ADA | 0
  Treatment boosted ADA | 0

35. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs): LPLV Analysis
Description: Adverse Event (AE) was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had a causal relationship with the treatment. TEAEs were defined as AEs that developed, worsened, or became serious during the treatment period (time from the first dose of study treatments up to 30 days after last dose of study treatments). An SAE was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability / incapacity, was a congenital anomaly/birth defect, was a medically important event.
Time Frame: From first dose of study treatment administration (Day 1) up to 30 days post last dose of study treatment administration, up to 349 weeks for Kd arm and 356 weeks for IKd arm (maximum duration of treatment exposure)
Population: Analysis was performed on safety population which included all who gave their informed consent and for whom there was confirmation of successful allocation of a randomization number by the IRT and received at least one dose or a part of a dose of the study treatments.
Measure: Count of Participants; unit: Participants
Groups:
- Isatuximab + Carfilzomib + Dexamethasone (IKd): Participants received isatuximab 10 mg/kg, IV infusion on Days 1, 8, 15 and 22 in Cycle 1, and then on Days 1 and Day 15 of each 28-day treatment cycle plus carfilzomib 20 mg/m^2, IV on Days 1, and 2 in Cycle 1, and then escalated to 56 mg/m^2 on Days 8, 9, 15 and 16 of Cycle 1 and then on Days 1, 2, 8, 9, 15 and 16 of each subsequent 28-day treatment cycle and dexamethasone 20 mg, PO or IV on Day 1, 2, 8, 9, 15, 16, 22 and 23 of each 28-day treatment cycle until disease progression or unacceptable adverse event or participant's decision to discontinue the study treatment or any other reason, whichever comes first (maximum exposure: 356 weeks).
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 122 | 177
Participants
  Any TEAE | 119 | 175
  Any treatment emergent SAE | 74 | 129

36. Primary Outcome: Progression Free Survival (PFS) As Determined by Independent Response Committee (IRC): Primary Analysis
Description: Time (in months) from randomization to date of 1st documentation of progressive disease (PD)/date of death from any cause, whichever comes 1st. If PD & death are not observed before cut-off date/date of initiation of further anti-myeloma treatment, PFS was censored at date of last valid disease assessment not showing PD performed prior to initiation of further anti-myeloma treatment/cut-off date, whichever comes 1st. PD(IMWG criteria):any 1 of following:Increase(inc) of >=25% in serum M-component from nadir; serum M component inc >=1 g/dL in 2 consecutive assessment, if starting M component >=5 g/dL; and/or inc of >=25% in urine M-component from nadir and/or development of new bone lesion/soft tissue extramedullary disease/inc >=50% from nadir in sum of perpendicular diameters of existing soft tissue extramedullary disease lesion if >1 lesion/ >=50% increase in longest diameter of previous soft tissue extramedullary disease lesion >1 cm in short axis. Estimated by Kaplan-Meier method.
Time Frame: From randomization until the primary analysis data cut-off date of 7 Feb 2020 (median duration of follow-up was 20.73 months)
Population: Analysis was performed on Intent to Treat (ITT) population that included all participants who gave their informed consent and for whom there was a confirmation of successful allocation of a randomization number by the interactive response technology (IRT).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
months | 19.15 [15.770 to NA] — Upper limit of the confidence interval could not be reached due to less number of participants with the events. | NA [NA to NA] — Median value and the upper and lower limit of the confidence interval could not be calculated because of less than 50% of the participants had PFS events.
Statistical Analysis 1: Comparison: Carfilzomib + Dexamethasone (Kd) vs Isatuximab + Carfilzomib + Dexamethasone (IKd); Statistical analysis for comparison of PFS between the Kd and IKd arms based on primary analysis; Test type: Superiority — For PFS, the nominal significance levels at primary analysis was determined using alpha-spending function in order to control overall 1-sided type 1 error at 2.5%. The 1-sided nominal significance level to declare overwhelming efficacy at primary analysis (103 PFS events) was 0.005. Because the median PFS was not reached at the primary analysis, it was described at the final analysis; p = 0.0007, Stratified Log-Rank test — One-sided p-value based on Stratified log-rank test. Threshold for statistical significance at 0.005; Stratified on number of prior lines of therapy (1 vs >1) & revised international staging system stage (I/II vs III vs not classified) as per IRT; Hazard Ratio (HR) = 0.531, 99% CI 2-sided [0.318 to 0.889] — Hazard Ratio was stratified on number of prior lines of therapy (1 vs. >1) and R-ISS stage (I or II vs. III vs. not classified) according to IRT

37. Primary Outcome: Progression Free Survival as Determined by Independent Response Committee: [Event Censored if Occurred >8 Weeks From Last Disease Assessment]: Primary Analysis
Description: Time (in months) from randomization to date of 1st PD documentation/death date, whichever is 1st. If PD & death not observed before cut-off date/date of further anti-myeloma treatment initiation, PFS censored at date of last valid disease assessment not showing PD performed prior to initiation of further anti-myeloma treatment/cut-off date, whichever was 1st. Progression/deaths occurring >8 weeks after last disease assessment censored at earliest date of last disease assessment without evidence of progression before initiation of new anti-myeloma treatment & cut-off date. PD (IMWG criteria): meeting any 1: Inc >=25% in Serum M-component from nadir; serum M component inc >=1 g/dL in 2 consecutive assessment, if starting M component >=5 g/dL; and/or inc >=25% in Urine M-component from nadir and/or development of new bone lesion/soft tissue extramedullary disease/inc >=50% from nadir in sum of perpendicular diameters of existing soft tissue extramedullary disease lesion >1 cm short axis.
Time Frame: as for outcome 1
Population: Analysis was performed on the ITT. Analysis was performed by Kaplan-Meier method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
months | 20.27 [15.770 to NA] — Upper limit of the confidence interval could not be reached due to less number of participants with the events. | NA [NA to NA] — Median value and the upper and lower limit of the confidence interval could not be calculated because of less than 50% of the participants had PFS events.
Statistical Analysis 1: Comparison: Carfilzomib + Dexamethasone (Kd) vs Isatuximab + Carfilzomib + Dexamethasone (IKd); Statistical analysis for comparison of PFS between the Kd and IKd arm based on primary analysis; Test type: Superiority — The 1-sided nominal significance level to declare overwhelming efficacy at primary analysis was 0.004. Because the median PFS was not reached at the primary analysis, it was described at the final analysis; p = 0.0016, Stratified Log-Rank test — One-sided p-value based on Stratified log-rank test. Threshold for statistical significance at 0.004; [statistical method as in outcome 36, analysis 1]; Hazard Ratio (HR) = 0.548, 99.2% CI 2-sided [0.317 to 0.948] — [estimate comment as in outcome 36, analysis 1]

38. Primary Outcome: Progression Free Survival as Determined by Independent Response Committee: Final Analysis
Description: PFS: time (in months) from randomization to date of first documentation of PD or date of death from any cause, whichever comes first. If PD and death are not observed before analysis cut-off date or date of initiation of further anti-myeloma treatment, PFS was censored at date of last valid disease assessment or analysis cut-off date, whichever comes first. PD as per IMWG criteria: any 1 of following: Inc of >=25% in Serum M-component from nadir; serum M component increase >=1 g/dL in 2 consecutive assessment, if starting M component was >=5 g/dL; and/or inc of >=25% in Urine M-component from nadir and/or development of new bone lesion/soft tissue extramedullary disease/inc >=50% from nadir in sum of perpendicular diameters of existing soft tissue extramedullary disease lesion if >1 lesion/ >=50% inc in longest diameter of previous soft tissue extramedullary disease lesion >1 cm in short axis. PFS estimated by Kaplan-Meier method.
Time Frame: From randomization until the final analysis data cut-off date of 14 January 2022 (the median duration of follow-up was 43.96 months)
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Carfilzomib + Dexamethasone (Kd): Participants received carfilzomib 20 milligrams per meter square (mg/m^2), intravenous (IV) infusion on Days 1, and 2 in Cycle 1, and then escalated to 56 mg/m^2 on Days 8, 9, 15 and 16 of Cycle 1 and then on Days 1, 2, 8, 9, 15 and 16 of each subsequent 28-day treatment cycle along with dexamethasone 20 milligrams (mg), orally (PO) or IV on Days 1, 2, 8, 9, 15, 16, 22 and 23 of each 28-day treatment cycle until disease progression or unacceptable adverse event or participant's decision to discontinue the study treatment or any other reason, whichever comes first (maximum exposure: 208 weeks).
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
months | 19.15 [15.770 to 25.035] | 35.65 [25.758 to 43.959]
Statistical Analysis 1: Comparison: Carfilzomib + Dexamethasone (Kd) vs Isatuximab + Carfilzomib + Dexamethasone (IKd); Test type: Superiority; Hazard Ratio (HR) = 0.576, 95.4% CI 2-sided [0.418 to 0.792] — [estimate comment as in outcome 36, analysis 1]

39. Primary Outcome: Progression Free Survival as Determined by Independent Response Committee [Event Censored if Occurred >8 Weeks From Last Disease Assessment]: Final Analysis
Description: Time (in months) from randomization to date of 1st documentation of PD/date of death from any cause, whichever comes 1st. If PD & death are not observed before cut-off date/date of initiation of further anti-myeloma treatment, PFS was censored at date of last valid disease assessment not showing PD/cut-off date, whichever comes 1st. Progressions/deaths occurring >8 weeks after last disease assessment were censored at earliest date of last valid disease assessment not showing PD before initiation of further anti-myeloma treatment & cut-off date. PD (per IMWG criteria): meeting any 1 criteria: Inc of >=25% in serum M-component from nadir; serum M component inc >=1 g/dL in 2 consecutive assessment, if starting M component was >=5 g/dL; and/or inc of >=25% in urine M-component from nadir and/or development of new bone lesion/soft tissue extramedullary disease/inc >=50% from nadir in sum of perpendicular diameters of existing soft tissue extramedullary disease lesion >1 cm in short axis.
Time Frame: as for outcome 4
Population: Analysis was performed on the ITT population. Analysis was performed by Kaplan-Meier method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
Number analyzed (Participants) | 123 | 179
months | 20.76 [16.164 to 28.189] | 41.66 [27.138 to NA] — Upper limit of the confidence interval could not be reached due to less number of participants with the events.
Statistical Analysis 1: Comparison: Carfilzomib + Dexamethasone (Kd) vs Isatuximab + Carfilzomib + Dexamethasone (IKd); Test type: Superiority; Hazard Ratio (HR) = 0.594, 95.4% CI 2-sided [0.424 to 0.832] — [estimate comment as in outcome 36, analysis 1]

ADVERSE EVENTS:
Time Frame: AE data and deaths were collected during the whole study. TEAEs that developed, worsened, or became serious during the treatment period were assessed from first dose of study treatment administration (Day 1) up to 30 days post last dose of study treatment administration, up to 349 weeks for Kd arm and 356 weeks for IKd arm (maximum duration of treatment exposure).
Description: AEs and SAEs were collected in safety population that included participants who received at least 1 dose or a part of a dose of the study treatments. All-Cause Mortality data collected during the study was assessed for all randomized participants. All-cause mortality (deaths) was assessed from randomization to the end of follow-up (FU) for each participant. Maximum time between randomization and those deaths observed in FU was up to approximately 297 weeks.
Arm/Group | Carfilzomib + Dexamethasone (Kd) | Isatuximab + Carfilzomib + Dexamethasone (IKd)
All-Cause Mortality (participants affected / at risk) | 59/123 | 83/179
Serious Adverse Events (participants affected / at risk) | 74/122 | 129/177
Other Adverse Events (participants affected / at risk) | 113/122 | 167/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carfilzomib + Dexamethasone (Kd) (N=122) | Isatuximab + Carfilzomib + Dexamethasone (IKd) (N=177)
Abdominal Abscess (Infections and infestations) | 1 (1) | 1 (1)
Abdominal Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Atypical Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial Infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3)
Bronchitis Pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 1 (2) | 5 (5)
Covid-19 Pneumonia (Infections and infestations) | 2 (2) | 4 (4)
Campylobacter Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (3) | 3 (3)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus Viraemia (Infections and infestations) | 0 (0) | 1 (2)
Device Related Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Escherichia Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (3) | 2 (2)
Gastroenteritis Salmonella (Infections and infestations) | 0 (0) | 1 (1)
H1n1 Influenza (Infections and infestations) | 0 (0) | 1 (1)
H3n2 Influenza (Infections and infestations) | 1 (1) | 0 (0)
Haematoma Infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 5 (5) | 2 (2)
Liver Abscess (Infections and infestations) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 6 (12) | 8 (8)
Lower Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 1 (1)
Metapneumovirus Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae Virus Infection (Infections and infestations) | 1 (1) | 2 (2)
Phlebitis Infective (Infections and infestations) | 1 (1) | 0 (0)
Pleurisy Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 17 (20) | 41 (54)
Pneumonia Influenzal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Legionella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Viral (Infections and infestations) | 0 (0) | 2 (2)
Pulmonary Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Respiratory Syncytial Virus Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 (0) | 3 (3)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 4 (4)
Salmonellosis (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 4 (4)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 6 (6)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary Tract Infection Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Vascular Device Infection (Infections and infestations) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 3 (3)
Visceral Leishmaniasis (Infections and infestations) | 0 (0) | 1 (2)
Anal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Breast Cancer Female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Large Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leptomeningeal Myelomatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Squamous Cell Carcinoma Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma Cell Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Second Primary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Normocytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Mineral Metabolism Disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Embolic Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial Mass (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 2 (2) | 1 (1)
Peripheral Nerve Paresis (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Deafness Neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 2 (3) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Aortic Valve Stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac Failure (Cardiac disorders) | 4 (5) | 5 (6)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure Chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Stenosis (Cardiac disorders) | 0 (0) | 2 (2)
Left Ventricular Failure (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 4 (4) | 3 (3)
Extremity Necrosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Venous Thrombosis Limb (Vascular disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Anal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis Ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 2 (2)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large Intestine Perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Diabetic Foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Chest Wall Haematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis Of Jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Sympathetic Posterior Cervical Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 5 (7) | 3 (3)
Calculus Urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrotic Syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Paraphimosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
Disease Progression (General disorders) | 2 (2) | 1 (1)
General Physical Health Deterioration (General disorders) | 1 (1) | 0 (0)
Injection Site Extravasation (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1)
Peripheral Swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 4 (4)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1)
Bone Marrow Plasmacyte Count Increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram T Wave Inversion (Investigations) | 0 (0) | 1 (1)
Grip Strength Decreased (Investigations) | 1 (1) | 0 (0)
Plasma Cells Increased (Investigations) | 1 (1) | 0 (0)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniofacial Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Multiple Injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Skin Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic Fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Traumatic Subarachnoid Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device Malfunction (Product Issues) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carfilzomib + Dexamethasone (Kd) (N=122) | Isatuximab + Carfilzomib + Dexamethasone (IKd) (N=177)
Bronchitis (Infections and infestations) | 14 (22) | 43 (71)
Covid-19 (Infections and infestations) | 2 (2) | 26 (31)
Conjunctivitis (Infections and infestations) | 9 (13) | 12 (13)
Gastroenteritis (Infections and infestations) | 7 (7) | 19 (23)
Influenza (Infections and infestations) | 13 (26) | 20 (27)
Lower Respiratory Tract Infection (Infections and infestations) | 8 (12) | 12 (16)
Nasopharyngitis (Infections and infestations) | 16 (30) | 36 (51)
Pneumonia (Infections and infestations) | 13 (21) | 18 (21)
Respiratory Tract Infection (Infections and infestations) | 7 (10) | 19 (49)
Rhinitis (Infections and infestations) | 3 (4) | 11 (18)
Sinusitis (Infections and infestations) | 5 (8) | 12 (20)
Upper Respiratory Tract Infection (Infections and infestations) | 32 (51) | 73 (189)
Urinary Tract Infection (Infections and infestations) | 11 (21) | 19 (32)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 9 (9)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 11 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (13) | 6 (6)
Decreased Appetite (Metabolism and nutrition disorders) | 5 (5) | 14 (18)
Anxiety (Psychiatric disorders) | 4 (5) | 15 (18)
Insomnia (Psychiatric disorders) | 30 (43) | 46 (54)
Dizziness (Nervous system disorders) | 7 (11) | 9 (13)
Headache (Nervous system disorders) | 22 (41) | 30 (43)
Peripheral Sensory Neuropathy (Nervous system disorders) | 16 (24) | 30 (36)
Cataract (Eye disorders) | 12 (13) | 31 (37)
Deep Vein Thrombosis (Vascular disorders) | 8 (9) | 8 (12)
Hypertension (Vascular disorders) | 42 (66) | 69 (109)
Superficial Vein Thrombosis (Vascular disorders) | 7 (12) | 10 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (30) | 41 (64)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 (42) | 54 (76)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 10 (13)
Abdominal Pain (Gastrointestinal disorders) | 9 (10) | 8 (12)
Abdominal Pain Upper (Gastrointestinal disorders) | 5 (5) | 9 (12)
Constipation (Gastrointestinal disorders) | 13 (17) | 25 (33)
Diarrhoea (Gastrointestinal disorders) | 38 (55) | 72 (134)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 17 (25)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 5 (5) | 12 (12)
Nausea (Gastrointestinal disorders) | 22 (35) | 39 (95)
Vomiting (Gastrointestinal disorders) | 13 (25) | 29 (49)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (12)
Rash (Skin and subcutaneous tissue disorders) | 9 (10) | 13 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (20) | 41 (64)
Back Pain (Musculoskeletal and connective tissue disorders) | 25 (34) | 43 (60)
Bone Pain (Musculoskeletal and connective tissue disorders) | 9 (12) | 14 (18)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 19 (26) | 28 (41)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 11 (14) | 6 (8)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 12 (12)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 17 (20) | 27 (36)
Asthenia (General disorders) | 21 (30) | 36 (71)
Fatigue (General disorders) | 25 (29) | 57 (82)
Influenza Like Illness (General disorders) | 5 (9) | 9 (13)
Non-Cardiac Chest Pain (General disorders) | 7 (8) | 11 (11)
Oedema Peripheral (General disorders) | 21 (31) | 30 (48)
Pyrexia (General disorders) | 21 (31) | 22 (34)
Weight Decreased (Investigations) | 1 (1) | 13 (13)
Accidental Overdose (Injury, poisoning and procedural complications) | 7 (8) | 17 (41)
Contusion (Injury, poisoning and procedural complications) | 6 (13) | 12 (19)
Fall (Injury, poisoning and procedural complications) | 12 (23) | 23 (31)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 4 (6) | 80 (122)
Limb Injury (Injury, poisoning and procedural complications) | 3 (5) | 11 (12)
Skin Laceration (Injury, poisoning and procedural complications) | 3 (7) | 11 (34)
Traumatic Fracture (Injury, poisoning and procedural complications) | 4 (5) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-11-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT03275285/Prot_004.pdf
  • Statistical Analysis Plan (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT03275285/SAP_005.pdf